CLINICAL TRIAL: NCT01681420
Title: Improving Blood Safety and HIV Testing in Brazil: a Randomized Controlled Trial
Brief Title: Improving Blood Safety and HIV Testing in Brazil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitalant Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 10849
Record Dates: First submitted 2012-02-29; First posted 2012-09-10 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: HIV; Herpes Simplex 2; Hepatitis C; Hepatitis B; Chagas Disease
Keywords: HIV counseling; Blood donor HIV testing; Brazil; Blood banks; Blood donors
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Chagas Disease | interventions — Blood Donation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Approved Intervention Counseling (Experimental): Approved blood donors randomized to intervention and choosing HIV counseling option with no donation.
  Interventions: Behavioral: HIV Counseling and Testing
- Approved Intervention Donation (Experimental): Approved blood donors randomized to intervention and choosing donation with no HIV counseling.
  Interventions: Behavioral: Blood Donation
- Deferred Intervention (Experimental): Deferred blood donors randomized to intervention with HIV counseling.
  Interventions: Behavioral: HIV Counseling and Testing

INTERVENTIONS:
Behavioral: HIV Counseling and Testing — HIV counseling and testing in lieu of blood donation.
  Arms: Approved Intervention Counseling; Deferred Intervention
Behavioral: Blood Donation — Blood donation without HIV counseling
  Arms: Approved Intervention Donation

SUMMARY:
Conduct a randomized controlled trial (RCT) to test the hypothesis that offering client-centered HIV counseling and testing (HCT) to blood donor candidates will reduce the risk of HIV contamination in the blood supply and also increase appropriate referrals to preventive and care services to persons in need in São Paulo, Brazil.

DETAILED DESCRIPTION:
Although all donated blood is screened for HIV antibodies, a residual risk of contamination persists due to the immunological window period before antibodies are detectable. Deferral of donors with behavioral risks for HIV is one means to reduce window period contamination; recruitment of voluntary donors from the community (versus family replacement donors) is held to be another. Contrary to expectation, a shift to community donors has not resulted in a decrease in HIV prevalence in units of blood collected by the investigators transfusion service. The investigators preliminary research indicates that some persons at elevated risk use donation as a means of testing for HIV. These test-seeking donors have high trust in the blood bank, do not know other places to receive testing, have low understanding of the immunological window period and believe it is acceptable to deny risk in order to be tested through donation. The test-seeking phenomenon may therefore threaten the safety of the blood supply. Test seeking at blood banks also ill serves persons who need risk reduction counseling because they cannot disclose their true behavior during the donation process and still be tested. Donors also have a low rate of return for test results and therefore do not receive confirmation or referrals to care.

To assess whether HCT at the time of donation will improve blood safety and address prevention and care needs, the investigators will randomize donor candidates to be offered this service on-site. As a biological marker for elevated risk for HIV, the investigators will compare the prevalence of HSV-2 among donors choosing testing to those choosing to donate when offered the choice (Aim 1). The impact of the intervention will be measured as an increase in persons receiving their test results, disclosure counseling and referrals (Aim 2). Secondary outcomes include differences in prevalence of transfusion-transmitted infections (HIV, HCV, HBV, syphilis, HTLV I/II, Chagas disease), donor motivations (e.g., test-seeking vs. altruism), donor deferral rates, use of confidential unit exclusion, satisfaction with procedures of the blood bank and volume of blood available for use. RCT results will provide rigorous evidence for or against the provision of on-site HCT as an effective means to improve blood safety and link individuals to needed health services.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects will be Portuguese-speaking persons age 18-65 years (determined by Brazilian law to be the age of donation), who present to donate blood at our center during the study period and who provide written informed consent.

Exclusion Criteria:

* All those not meeting inclusion criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11900 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
HSV-2 Prevalence in Blood Donors | Up to three years.
  As a biological marker for elevated risk for HIV, we will compare the prevalence of HSV-2 among donors choosing testing to those choosing to donate when offered the choice.
Intervention Impact in Blood Donors | Up to three years.
  The impact of the intervention will be measured as an increase in persons receiving their test results, disclosure counseling and referrals.

SECONDARY OUTCOMES:
Prevalence of Transfusion-Transmitted Infections in Blood Donors | Up to three years.
  Differences in prevalence of transfusion-transmitted infections (HIV, HCV, HBV, syphilis, HTLV I/II, Chagas disease) between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Thelma T. Goncalez, MD, PhD, Principal Investigator — Vitalant Research Institute
Locations (1):
- Fundação Pró-sangue Hemocentro de São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Goncalez TT, Blatyta PF, Santos FM, Montebello S, Esposti SP, Hangai FN, Salles NA, Mendrone A, Truong HM, Sabino EC, McFarland W. Does offering human immunodeficiency virus testing at the time of blood donation reduce transfusion transmission risk and increase disclosure counseling? Results of a randomized controlled trial, Sao Paulo, Brazil. Transfusion. 2015 Jun;55(6):1214-22. doi: 10.1111/trf.13009. Epub 2015 Feb 3. PMID 25646883